CLINICAL TRIAL: NCT06908915
Title: Long Pulse 1064 nm Nd:YAG Laser in the Treatment of Erythematotelangiectatic Rosacea and Other Erythematous Telangiectatic Facial Conditions
Acronym: Nd:YAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Dindar Sharif Qurtas, Asst Professor, Hawler Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KHCMS: 12/241-2023
Record Dates: First submitted 2024-12-28; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Rosacea, Erythematotelangiectatic
Keywords: Nd:YAG laser
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Definition: rosacea patients. Limit: 30 patients (Experimental): Patients with rosacea received treatment with Nd:YAG laser with spot size: 5mm, fluence: 4.07 J/Cm2, energy: 800 mJ and frequency: 5 Hz. About 2-3 passes performed in each treatment session. Up to four sessions were performed for each patient with 2 weeks interval
  Interventions: Device: Nd:YAG laser 1064 nm

INTERVENTIONS:
Device: Nd:YAG laser 1064 nm — The entire face of each patient with rosacea was treated with long-pulse 1064nm Nd:YAG laser. The parameters that been used were spot size: 5mm, fluence: 4.07 J/Cm2, energy: 800 mJ and frequency: 5 Hz. About 2-3 passes performed in each treatment session. Up to four sessions were performed for each patient with 2 weeks interval.

SUMMARY:
The goal of this clinical study is to assess the effectiveness of Nd:YAG laser 1064 nm in the long pulse mode in the treatment of signs of rosacea including the erythema of the face and telangiectasia. The used parameter of this laser was of very low energy (spot size: 5mm, fluence: 4.07 J/Cm2, energy: 800 millijoules (mJ) and frequency: 5 Hz. About 2-3 passes performed in each treatment session. Up to four sessions were performed for each patient with 2 weeks interval) and also its was expected to have minimal adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Patient with rosacea (erythemato-telangiectatic type)

Exclusion Criteria:

* Other clinical types of rosacea
* Pregnancy and lactation in females
* History of malignancies
* History of photosensitivity
* History of any other modalities of treatment of rosacea over last 6 months

Ages: 32 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Changes in erythema of face of patients with rosacea been treated by ND:YAG laser 1064 nm long pulse width by using clinician erythema scale (CEA) | Three months
  Erythema was graded from 0 to 4 using clinician erythema assessment scale (CEA). The score 0 is the lowest score of erythema and score 4 means the highest severity of erythema of the skin

CONTACTS AND LOCATIONS:
Locations (1):
- Hawler Medical University, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: Yes